CLINICAL TRIAL: NCT04537390
Title: Anti-mullerian Hormone Levels in Healthy Females
Acronym: AMH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erin Rowell (Other)
Collaborators: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Sponsor-Investigator, Erin Rowell, Director, Ann & Robert H Lurie Children's Hospital of Chicago
Organization: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-610
Record Dates: First submitted 2020-08-28; First posted 2020-09-03 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Healthy
Keywords: AMH

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Blood sample collection (Other): Blood samples are collected for diagnostically assessing how the blood AMH levels correspond to a female's reproductive development
  Interventions: Diagnostic Test: Blood sample collection

INTERVENTIONS:
Diagnostic Test: Blood sample collection — Blood samples are collected for diagnostically assessing how the blood AMH levels correspond to a female's reproductive development

SUMMARY:
The purpose of this study is to have a better understanding of the normal blood levels of AMH in females from 0-18 years of age and how the blood AMH levels correspond to a female's reproductive development.

DETAILED DESCRIPTION:
Anti-mullerian hormone (AMH) is a chemical in the body that is found in the blood that can estimate the ability of a female to have her own children. It is widely used in adult female cancer patients to predict the onset of menopause and/or the inability to have children that can be associated with chemotherapy and/or radiation treatment. Normal blood levels of AMH are better understood in adults than in children and adolescents. The purpose of this study is to have a better understanding of the normal blood levels of AMH in females from 0-18 years of age and how the blood AMH levels correspond to a female's reproductive development. With a better understanding of normal AMH levels in children, we may be able to better assess a girl's risk of not being able to have children if she is a cancer patient, and may be able to offer her and her family options to increase the chances of having her own children.

ELIGIBILITY:
Inclusion Criteria:

1. Pre- and post-pubertal females
2. Ages 0-18 years old
3. Tanner Stage I- V
4. Undergoing routine outpatient surgical procedure

   1. Hernia repair (inguinal, umbilical, epigastric)
   2. Excision of benign mass
   3. laparoscopic cholecystectomy

Exclusion Criteria:

1. Previous diagnosis of an illness associated with premature ovarian failure (Turner's syndrome, Fragile X permutation carrier) or endocrine disorder associated with irregular menstrual cycles (Cushing's disease, poorly-controlled Thyroid disease, hyperprolactinemia, polycystic ovary syndrome, and congenital adrenal hyperplasia) or insulin-dependent diabetes mellitus or autoimmune disorders
2. Previous diagnosis of any malignancy or any history of systemic/local chemotherapy, radiation therapy, or stem-cell transplant.
3. Previous surgical excision of one ovary or both ovaries
4. Pregnant females
5. All inpatient surgical patients
6. Undergoing non-routine outpatient surgical procedures

   1. Central venous catheter placement
   2. Supprelin insertion/removal
   3. Breast mass excision
   4. Gastrostomy tube insertion

Max Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2016-07-19 (Actual); Primary Completion 2030-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Anti-mullerian Hormone Levels in Healthy Females | 3 Years
  The primary outcome measure is to get a better understanding of the normal AMH levels in children (girls aged 0-18 years) in order to better assess a girl's risk of not being able to have children if she is a cancer patient, and in offering her and her family options to increase the chances of having her own children

CONTACTS AND LOCATIONS:
Overall Officials: Erin Rowell, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No